CLINICAL TRIAL: NCT07119112
Title: Evaluation of a Novel Drain Stripping Device for Reducing Surgical Drain Complications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rob B. Hill, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-006697
Record Dates: First submitted 2025-07-18; First posted 2025-08-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Surgical Drain; Abdominal Surgery Patients; Drains
Keywords: Surgical Drain; Drain Tube Clearance; Drain Tube Occlusion; Drain Clearance Device
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: We are comparing single group device user(s) to standard of care model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain device user(s) (Experimental): Study participants whose caregivers are utilizing the drain device to clear surgical drain tubing.
  Interventions: Device: Surgical drain stripping device
- Control (Other): Study participants whose caregivers use the current standard of care for surgical drain tube stripping.
  Interventions: Other: Standard of Care (Investigator Choice)

INTERVENTIONS:
Device: Surgical drain stripping device — We have developed a device to fully compress the surgical drain tubing without compromising the integrity of the tubing to clear the drain fluid/debris more effectively than the current standard of care.
  Arms: Drain device user(s)
Other: Standard of Care (Investigator Choice) — Current standard of care for surgical drain tube stripping involves running fingertips down the length of the tubing compressing the drain tubing to clear fluid/debris.
  Arms: Control

SUMMARY:
The purpose of this research is to evaluate how well a novel surgical site drain tube clearing device works, and how easy it is for care staff to use.

DETAILED DESCRIPTION:
The purpose of this research is to gather information on the ease of use, effectiveness, and potential ability to reduce post-surgical drain complications of a drain stripping device which was developed and made here at the Mayo Clinic. The device has been patented and has been tested in laboratory conditions, but it has not yet been evaluated by the FDA or cleared for marketing yet since it is a device that poses minimal risk to patients. The device is a plastic clamp which is used to move fluid through the drain tubing to keep the tubing clear and free flowing. The current method (standard of care) for doing this simply involves running fingers down the tubing to drain the fluid, which can be inadequate and sometimes physically challenging. The primary goal of the study is to get feedback from nurses using the device in a clinical setting. There are approximately 80 nurses working the hospital unit which cares for patients who may have a post-surgical drain emplaced. We will gather their feedback via an anonymous survey which will be available to the nurses on the Mayo Clinic Intranet. Secondary goals of the study attempt to ascertain the potential effect of device use upon patient outcomes. Inadequate draining of surgical site fluid can sometimes create the need for additional interventions, including surgical revisions. The drain stripping device used in this study, has been developed to address these issues. Preliminary bench testing in laboratory conditions has not indicated any reason to believe that use of the device to clear surgical drain tubing poses any greater (or even different) risk to patients than the current standard of care (using bare fingers). Patients are routinely sent home with one or more surgical drains which are cleared by the patient using the current standard of care. Therefore, there is no safety related need to start with a small number of study subjects as is typical for an initial trial; and since this is not a device or drug which would be likely to show obvious benefit within a small cohort, we are seeking data regarding potential effect of study device upon patient outcomes from 420 study subject encounters (210 in each arm - device use versus current standard of care), as opposed to the small numbers of subjects usually seen in initial clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older, with no maximum age limit.
* Patients undergoing surgical procedures that require the placement of Jackson-Pratt drains within the abdominal cavity.
* Patients who are able to provide informed consent for participation in the study.
* Mayo Clinic RNs caring for patients with post-surgical drains placed.

Exclusion Criteria:

* Patients under the age of 18.
* Patients who do not have Jackson-Pratt drains placed post-operatively.
* Patients with drains placed in locations other than the abdominal cavity.
* Patients with known allergies or contraindications to the materials used in the drain stripping device.
* Patients who are unable to provide informed consent due to cognitive impairments or any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Assess Ease of Use and Device Functionality Via Anonymous Survey | 1 year
  Gather and analyze feedback from nurses regarding the ease of device use and the ability of the device to clear surgical drain tubing in the clinical setting via an anonymous survey which nurses may access within the Mayo Clinic intranet.

SECONDARY OUTCOMES:
Assess Effect Study Device May Have Upon Duration of Surgical Drain Placement | 1 year
  Compare device use and standard of care group of study subjects for the amount of time their surgical drains remain in place to assess the potential ability of the surgical drain stripping device to reduce the time needed for a surgical drain to remain in place (in situ).
Assess Whether Device Reduces Surgical Drain Complications | 1 year
  Compare clinical outcomes between device use and standard of care study subjects to assess whether or not the surgical drain tube stripping device leads to fewer drain associated post operative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hill, APRN,CNP,MSN, Principal Investigator — Mayo Clinic; Michael Thorn, APRN,CNP,MSN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
The primary study goal involves collecting device use feedback via an anonymous survey, and the secondary goals involve collecting and analyzing collective data. There would be no benefit to anyone to share individual study subject data, and we would not want to consider adding a patient privacy risk factor without obvious benefit.